CLINICAL TRIAL: NCT06361472
Title: A Single-Center, Investigator-Blinded, Randomized, 4-Week, Parallel-Group, Superiority Study Comparing Contextual Factors-Enriched Standard Care Versus Standard Care Only for Patients with Mechanical Neck Pain (ContextualizAR Trial)
Brief Title: Contextual Factors-Enriched Standard Care on Mechanical Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de la Matanza (Other)
Responsible Party: Principal Investigator, Mauro Federico Andreu, Prof. Mauro Federico Andreu, PhD, Universidad Nacional de la Matanza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11695
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Neck Pain
Keywords: neck pain; functional status; contextual factors; placebo; randomized controlled trial
MeSH Terms: conditions — Neck Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The ContextualizAR trial is designed as a two-arm, randomized, controlled, and blinded assessor superiority trial conducted at a single center. Patients will be allocated to one of two groups: a CFs+SC group and the SC group.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, blinding of both therapists and patients will not be feasible. However, to uphold the scientific validity of the study, specific descriptors and methodological details, such as terms like "placebo" or "CFs," have been intentionally excluded from the consent disclosure. To prevent any potential bias in participants' perceptions, information regarding the potential involvement of CFs in outcomes will not be provided. Instead, participants will be informed that the study aims to assess changes resulting from standard treatment for MNP. The person in charge of data statistical analysis (FV) and the evaluators who will assess all participants' pre- and post-intervention assessments (MLL and AR) will be blinded to the allocated intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care (SC) (Active Comparator): Treatment will be carried out based on the mechanical neck pain clinical practice guideline. Physiotherapists treating this group of patients will avoid enhancing the contextual factors mentioned in the intervention group.
  Interventions: Other: Standard Care
- Contextual Factors-Enriched Standard Care (CFs+SC) (Experimental): Treatment will be carried out based on the mechanical neck pain clinical practice guideline. Additionally, Contextual Factors, which include physical, psychological, and social elements involved in the clinical encounter between the patient and the physiotherapist, will be deliberately enhanced in this group.
  Interventions: Other: Standard Care; Behavioral: Contextual Factors

INTERVENTIONS:
Other: Standard Care — Standard Care includes exercises, mobilization, manual therapy, education, and Neck Wellness Home Care Guide (NWHCG). The rehabilitation program is based on current clinical practice guidelines aimed at reducing neck pain, improving range of motion, enhancing functionality, and promoting physical activity motivation. Each patient will receive active exercises and manual therapy techniques. Educational components will cover pain science, physical activity benefits, and return to normal activities , supplemented by a NWHCG. Treatment sessions will be conducted, featuring a one-to-one interaction between the participant and the physiotherapist. It will last 4 weeks, with two sessions per week, 45 minutes/session (8 treatment sessions).
  Other Names: SC
Behavioral: Contextual Factors — Bundle of contextual factors divided into three categories: professional, treatment, and healthcare setting features. Regarding the professional contextual factors, they include reputation, appearance, and positive attitudes. The treatment contextual factors encompass positive attitudes, verbal communication, non-verbal communication, empathetic therapeutic alliance, therapeutic touch, and the use of a mirror to show the patient what is being performed. Finally, the healthcare setting contextual factors feature a comfortable setting, adequate environmental conditions, and appropriate design.
  Other Names: CFs
  Arms: Contextual Factors-Enriched Standard Care (CFs+SC)

SUMMARY:
The primary purpose of this study will be to determine if a CFs-Enriched Standard Care approach is an effective treatment for mechanical neck pain in terms of reducing pain and improving function. We hypothesize that a 4-week CFs-Enriched Standard Care approach will be superior to Standard Care alone in terms of patient-reported disability and pain, with measurements conducted using the Northwick Park Neck Pain Questionnaire and the Numeric Pain Rating Scale, respectively.

This will be an assessor-blinded, 2-group (1:1) randomized clinical trial aiming to enroll 94 participants with neck pain persisting for more than 4 weeks. Both groups will undergo 4 weeks of standard care twice weekly, following established clinical practice guidelines. In the intervention group, CFs will be enhanced, encompassing the physical, psychological, and social elements inherent in the clinical encounter, based on existing evidence.

The primary outcomes will encompass changes in Pain and Disability after 4 weeks of treatment, with a follow-up reassessment at week 12 post-treatment. Secondary outcomes will include changes in Active Range of Motion, Global Rating of Change, and Satisfaction with treatment. The change between groups after treatment and at the 12-week follow-up will be reported for all outcomes, considering the difference from scores recorded at baseline.

DETAILED DESCRIPTION:
The primary aim of this study is to determine if a Contextual Factors-Enriched Standard Care (CFs+SC) approach is an effective treatment for MNP in terms of reducing pain and improving function. We hypothesize that a 4-week Contextual Factors-Enriched Standard Care will be superior to Standard Care alone in terms of patient-reported disability and pain, with measurements conducted using the Argentine version of the Northwick Park Neck Pain Questionnaire (NPQ-AR) and the Numerical Pain Rating Scale (NPRS), respectively.

The secondary aims are:

* To determine whether CFs+SC is more effective than SC in terms of active range of motion (ROM) enhancement, global perceived effect (GROC), and satisfaction with treatment after the 4-week intervention.
* To determine if a CFs+SC approach is effective in treating MNP in terms of disability improvement, pain reduction, active ROM enhancement, global perceived effect (GROC), and satisfaction with treatment 12 weeks after a 4-week treatment plan.
* To explore differences in treatment credibility and expectations between the CFs+SC group and the SC group at both the 2-week and 4-week intervals.
* To investigate whether individuals identified with at least one negative psychosocial condition (such as anxiety, fear of movement, stress, catastrophizing, and depression) will experience greater benefits from the CFs+SC intervention compared to those without negative psychosocial conditions.

Consecutive patients meeting all inclusion criteria and none of the exclusion criteria will be randomly assigned in a 1:1 ratio to either the CFs+SC group or the SC alone group. Randomization will employ a blocked design with variable block lengths (2:4) and will be stratified based on baseline pain ('mild-moderate' or 'severe,' determined by whether they report between 3 and 7 points or ≥ 8 points on the baseline NPRS, respectively) and participants' expectations ('high' or 'low') regarding the effectiveness of standard care treatment.

The randomization process will be generated and conducted by SS and PP, who will not be involved in data analysis or patient enrollment. The website www.randomization.com will be used for this process. To maintain allocation concealment during the study, sequential, numbered, and sealed opaque envelopes will be utilized. Patients will be allocated to one of two groups: a CFs+SC group and the SC group. Due to the nature of the study, blinding of both therapists and patients will not be feasible. The person in charge of data statistical analysis (FV) and the evaluators who will assess all participants' pre- and post-intervention assessments (MLL and AR) will be blinded to the allocated intervention.

Both groups will undergo 4 weeks of standard care twice weekly following established clinical practice guidelines, and including exercises, mobilization, manual therapy, education, and a neck wellness home care guide. In the intervention group, CFs will be enhanced, encompassing the physical, psychological, and social elements inherent in the clinical encounter, based on existing evidence.

At the onset of treatment, patients will receive a schedule outlining the dates of the next 8 visits. One day before each session, an individual not involved in the study will send a text message (SMS) reminder. Should a scheduled session be missed, it will be rescheduled. However, patients who miss two consecutive scheduled sessions will be deemed dropouts and analyzed using the intention-to-treat (ITT) approach, with the last observed value taken into consideration. Additionally, participants will be asked to refrain from undergoing any other treatments until the end of the 12-week follow-up period. During this period, participants are only permitted to adhere to the NWHCG. If a participant reports undergoing any other treatments, they will be considered as dropouts and analyzed using the ITT approach.

Physiotherapists will undergo a comprehensive training program comprising 8 hours of formal instruction, tailored to provide the necessary skills and proficiency for both therapeutic contexts under investigation. To ensure treatment fidelity, a Manual of Treatment (MOT) was developed. Therapist adherence to the MOT will be evaluated through self-assessment ratings provided by the therapists themselves. After each session, therapists will rate their adherence to the manual using a form specifically designed for this study. Additionally, monthly audits will assess compliance with the MOT, and frequent meetings with providers will be held to mitigate any deviations in provider adherence to the MOT, ensuring its consistency over time.

The sample size for this study was determined using a linear mixed effects model to account for within-subject correlation arising from repeated measures over time. The model includes fixed effects, such as treatment group (CF+SC and SC groups), and time points (baseline, 4 weeks, and 12 weeks after treatment), along with the interaction between treatment group and time to assess potential changes in treatment effects over time. Random effects for individual subjects were also included to address repeated measures within the same subjects. Based on an assumed medium effect size (f2 = 0.15), 80% power, and a significance level of 0.05 (two-tailed), the estimated sample size required for this study was calculated to be 85 subjects. To accommodate a projected dropout rate of 10%, the sample size was adjusted, resulting in a final target sample size of 94 subjects (47 participants per group).

Outcomes will be analyzed on an ITT basis, with reporting of sample characteristics and descriptive statistics. Linear mixed models will be used for primary analysis to verify the differences between the average effects of interventions (CFs+SC and SC) in reassessments carried out 4 weeks after random allocation and 12 weeks after treatment. The differences between groups will be calculated by interaction terms of groups versus time. All statistical procedures will be performed using SPSS, developed by SPSS Inc., Chicago, IL, USA.

Trial procedures and evaluations will be conducted by trained personnel (MLL, AR, MM, GD, and FR) using paper-based Case Report Forms (CRFs), with implemented quality control measures. Subsequently, MM, GD, and FR will enter the data into an electronic database using MAWE® Data Collection Tools (www.mawetools.com). An independent data monitoring committee (MFA, SS, FV, and PP) will oversee the entire data collection process to ensure its quality and integrity. Monitoring of the study will be overseen by MFA and FV, encompassing verification of adherence to predefined inclusion and exclusion criteria, monitoring overall study progress, and ensuring accurate data recording in CRFs. Auditing responsibilities will be carried out weekly by the principal investigator to ensure completeness and accuracy across critical study components, including participant consent forms, paper forms, and recruitment rates.

The trial will be conducted in compliance with the principles of the Declaration of Helsinki, Good Clinical Practice, and all applicable regulatory requirements. Ethical approval has been obtained from the Institutional Review Board (IRB) (#11695, approved on 15/03/2024). The principal investigator and researchers affirm no financial or other competing interests. Access to final trial data will be provided to designated individuals and authorized personnel, with any contractual restrictions transparently disclosed. Upon trial completion, results will be published in peer-reviewed journals, following authorship guidelines established by the ICMJE and CRediT framework.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18.
* Neck pain for more than 4 weeks without signs or symptoms suggestive of major structural pathology.
* Read, write, and understand the Spanish language.
* Signed consent form.

Exclusion Criteria:

* Numeric Pain Reporting Scale (NPRS) < 3 points (to ensure the exclusion of patients with minor disorders).
* Northwick Park Neck Pain Questionnaire (NPQ) < 10 points (to ensure the exclusion of patients with minor disorders).
* History of cervical spine trauma, fracture, or surgical procedures.
* Signs and symptoms of cervical myelopathy and/or cervical radiculopathy (to rule out cervical radicular pain, the Spurling Test, the Upper Limb Tension Test for the median nerve, and the Traction/Distraction test will be used).
* Red flags or serious pathologies, such as malignancy, inflammatory or rheumatic diseases, infections, and vascular conditions like cervical artery insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Neck Pain Intensity | 4 weeks and 12 weeks after end of treatment
  Neck pain intensity will be measured using a Numerical Pain Rating Scale (NPRS) composed of an 11-point scale, ranging from 0 ("no pain") to 10 ("the "worst pain imaginable") (Hawker et al., 2011; Kahl & Cleland, 2005). In this study patients will be asked about their average pain intensity in the last 7 days (Jensen 1999).
Neck Disability | 4 weeks and 12 weeks after end of treatment
  Neck disability will be measured using the Argentinian version of the Northwick Park Neck Pain Questionnaire (NPQ-AR) (Aguirre et al., 2013). The questionnaire has 9 items relating to daily activities (personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation) and cervical spine pain. Each item is scored from 0 to 4, the total score is 36; higher scores represent higher pain or disability.

SECONDARY OUTCOMES:
Active Range of Movement | 4 weeks and 12 weeks after end of treatment
  AROM will be measured with the "clinometer" iPhone and/or Android app as described by Monreal (2021): Cervical flexion, extension, and lateral flexion measurements will be conducted with participants in a seated position
Global Rating of Change | 4 weeks and 12 weeks after end of treatment
  The GROC is designed to quantify a patient's improvement or deterioration over time. It requires the subject to evaluate his or her current health status and compare it to his or her previous condition (Kamper et al., 2009). To assess this construct the 10th question of the NPQ will be used. This item has 5 categories: ''much worse'', "Slightly worse", "The same", "Slightly better" and ''much better'' (Aguirre 2013).
Satisfaction with treatment | 4 weeks and 12 weeks after end of treatment
  Overall treatment satisfaction will be evaluated with question number 11 of the MedRisk questionnaire. (Beattie 2005) Patient will score from 1 (strongly disagree) to 5 (strongly agree), the following sentence: "Overall, I am completely satisfied with the services I receive from my therapist" (Beattie 2005).
Expectations | At baseline, at the end of week 2 (session 5), and at the conclusion of week 4 (session 9).
  Four questions, each corresponding to the specific intervention in the therapeutic plan (active exercises, manual therapy, education, and 'Neck Wellness Home Care Guide'), will be used to assess participants' expectations for the effectiveness of treatment. Participants will respond to the statement: 'I believe [intervention] will significantly help to improve this episode of my neck pain,' using a five-point scale: 'definitely agree,' 'agree,' 'neutral,' 'disagree,' and 'definitely disagree,' with 'neutral' representing the midpoint response (Bishop et al., 2013b).
Credibility | At baseline, at the end of week 2 (session 5), and at the conclusion of week 4 (session 9).
  The credibility regarding the treatment will be evaluated by the first three questions of the Credibility/Expectancy Questionnaire (Devilly & Borkovec, 2000). The three items addressing therapy credibility relate to: 1) the extent to which the treatment appears logical, 2) the extent to which the treatment appears useful, 3) the confidence with which the patient would recommend the treatment to a friend having the same problem.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro F Andreu, PhD, Principal Investigator — Universidad Nacional de la Matanza
Locations (1):
- Hospital Donación Francisco Santojanni, Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossettini G, Carlino E, Testa M. Clinical relevance of contextual factors as triggers of placebo and nocebo effects in musculoskeletal pain. BMC Musculoskelet Disord. 2018 Jan 22;19(1):27. doi: 10.1186/s12891-018-1943-8. PMID 29357856
- [Background] Kamper SJ. Engaging With Research: Linking Evidence With Practice. J Orthop Sports Phys Ther. 2018 Jun;48(6):512-513. doi: 10.2519/jospt.2018.0701. PMID 29852839
- [Background] Cook CE, Bailliard A, Bent JA, Bialosky JE, Carlino E, Colloca L, Esteves JE, Newell D, Palese A, Reed WR, Vilardaga JP, Rossettini G. An international consensus definition for contextual factors: findings from a nominal group technique. Front Psychol. 2023 Jul 3;14:1178560. doi: 10.3389/fpsyg.2023.1178560. eCollection 2023. PMID 37465492
- [Background] Testa M, Rossettini G. Enhance placebo, avoid nocebo: How contextual factors affect physiotherapy outcomes. Man Ther. 2016 Aug;24:65-74. doi: 10.1016/j.math.2016.04.006. Epub 2016 Apr 20. PMID 27133031
- [Background] Di Blasi Z, Harkness E, Ernst E, Georgiou A, Kleijnen J. Influence of context effects on health outcomes: a systematic review. Lancet. 2001 Mar 10;357(9258):757-62. doi: 10.1016/s0140-6736(00)04169-6. PMID 11253970
- [Background] Rossettini G, Camerone EM, Carlino E, Benedetti F, Testa M. Context matters: the psychoneurobiological determinants of placebo, nocebo and context-related effects in physiotherapy. Arch Physiother. 2020 Jun 11;10:11. doi: 10.1186/s40945-020-00082-y. eCollection 2020. PMID 32537245
- [Background] O'Keeffe M, Cullinane P, Hurley J, Leahy I, Bunzli S, O'Sullivan PB, O'Sullivan K. What Influences Patient-Therapist Interactions in Musculoskeletal Physical Therapy? Qualitative Systematic Review and Meta-Synthesis. Phys Ther. 2016 May;96(5):609-22. doi: 10.2522/ptj.20150240. Epub 2015 Oct 1. PMID 26427530
- [Background] Hush JM, Cameron K, Mackey M. Patient satisfaction with musculoskeletal physical therapy care: a systematic review. Phys Ther. 2011 Jan;91(1):25-36. doi: 10.2522/ptj.20100061. Epub 2010 Nov 11. PMID 21071504
- [Background] Andreu M, Policastro PO. ¿Por qué son importantes los factores contextuales en el abordaje kinésico? [Why are contextual factors important in the physical therapy approach?]. AJRPT. 2020;2(3):1-3. doi: 10.58172/ajrpt.v2i3.125
- [Background] Bialosky JE, George SZ, Bishop MD. How spinal manipulative therapy works: why ask why? J Orthop Sports Phys Ther. 2008 Jun;38(6):293-5. doi: 10.2519/jospt.2008.0118. Epub 2008 May 27. No abstract available. PMID 18515964
- [Background] Fuentes J, Armijo-Olivo S, Funabashi M, Miciak M, Dick B, Warren S, Rashiq S, Magee DJ, Gross DP. Enhanced therapeutic alliance modulates pain intensity and muscle pain sensitivity in patients with chronic low back pain: an experimental controlled study. Phys Ther. 2014 Apr;94(4):477-89. doi: 10.2522/ptj.20130118. Epub 2013 Dec 5. PMID 24309616
- [Background] Hu T, Long Y, Wei L, Zheng Y, Tong Y, Yuan M, Liu C, Wang X, Lin Y, Guo Q, Huang J, Du L. The Underappreciated Placebo Effects and Responses in Randomized Controlled Trials on Neck Pain: A Systematic Review With Meta-analysis. Arch Phys Med Rehabil. 2023 Jul;104(7):1124-1131. doi: 10.1016/j.apmr.2022.10.013. Epub 2022 Nov 20. PMID 36417969
- [Background] Pedersen JR, Strijkers R, Gerger H, Koes B, Chiarotto A. Clinical improvements due to specific effects and placebo effects in conservative interventions and changes observed with no treatment in randomized controlled trials of patients with chronic nonspecific low back pain: a systematic review and meta-analysis. Pain. 2024 Jun 1;165(6):1217-1232. doi: 10.1097/j.pain.0000000000003151. Epub 2024 Jan 10. PMID 38198235
- [Background] Tsutsumi Y, Tsujimoto Y, Tajika A, Omae K, Fujii T, Onishi A, Kataoka Y, Katsura M, Noma H, Sahker E, Ostinelli EG, Furukawa TA. Proportion attributable to contextual effects in general medicine: a meta-epidemiological study based on Cochrane reviews. BMJ Evid Based Med. 2023 Feb;28(1):40-47. doi: 10.1136/bmjebm-2021-111861. Epub 2022 Jul 19. PMID 35853683
- [Background] Miciak M, Gross DP, Joyce A. A review of the psychotherapeutic 'common factors' model and its application in physical therapy: the need to consider general effects in physical therapy practice. Scand J Caring Sci. 2012 Jun;26(2):394-403. doi: 10.1111/j.1471-6712.2011.00923.x. Epub 2011 Sep 14. PMID 21913950
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Childs JD, Cleland JA, Elliott JM, Teyhen DS, Wainner RS, Whitman JM, Sopky BJ, Godges JJ, Flynn TW; American Physical Therapy Association. Neck pain: Clinical practice guidelines linked to the International Classification of Functioning, Disability, and Health from the Orthopedic Section of the American Physical Therapy Association. J Orthop Sports Phys Ther. 2008 Sep;38(9):A1-A34. doi: 10.2519/jospt.2008.0303. Epub 2008 Sep 1. PMID 18758050
- [Background] Bier JD, Scholten-Peeters WGM, Staal JB, Pool J, van Tulder MW, Beekman E, Knoop J, Meerhoff G, Verhagen AP. Clinical Practice Guideline for Physical Therapy Assessment and Treatment in Patients With Nonspecific Neck Pain. Phys Ther. 2018 Mar 1;98(3):162-171. doi: 10.1093/ptj/pzx118. PMID 29228289
- [Background] Aguirre MV, Rodriguez MG, Clarett M, Iribarne JI, Martinez M, Battistotti R, Lopez de Arcaute AS, Adarves R, Orsini E. [Cultural adaptation and Argentine validation of the Northwick Park Neck Pain Questionnaire in the hospitals of the Autonomous City of Buenos Aires]. Rev Fac Cien Med Univ Nac Cordoba. 2013;70(2):76-82. Spanish. PMID 24067591
- [Background] Monreal C, Luinstra L, Larkins L, May J. Validity and Intrarater Reliability Using a Smartphone Clinometer Application to Measure Active Cervical Range of Motion Including Rotation Measurements in Supine. J Sport Rehabil. 2020 Sep 15;30(4):680-684. doi: 10.1123/jsr.2019-0422. PMID 32932236
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Beattie P, Turner C, Dowda M, Michener L, Nelson R. The MedRisk Instrument for Measuring Patient Satisfaction With Physical Therapy Care: a psychometric analysis. J Orthop Sports Phys Ther. 2005 Jan;35(1):24-32. doi: 10.2519/jospt.2005.35.1.24. PMID 15754601
- [Background] Bishop MD, Mintken PE, Bialosky JE, Cleland JA. Patient expectations of benefit from interventions for neck pain and resulting influence on outcomes. J Orthop Sports Phys Ther. 2013;43(7):457-65. doi: 10.2519/jospt.2013.4492. Epub 2013 Mar 18. PMID 23508341
- [Background] Okezue OC, Nwafor GC, Ezeukwu OA, et al. Adherence to Home Exercise Programmes and its Associated Factors among Patients Receiving Physiotherapy. ClinHealthPromot [Internet]. 2019 May 31 [cited 2024 Jan. 9];9(1):7-14. Available from: https://clinhealthpromot.org/index.php/clinhp/article/view/clinhp19003
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Cook CE, O'Halloran B, McDevitt A, Keefe FJ. Specific and shared mechanisms associated with treatment for chronic neck pain: study protocol for the SS-MECH trial. J Man Manip Ther. 2024 Feb;32(1):85-95. doi: 10.1080/10669817.2023.2267391. Epub 2024 Jan 16. PMID 37819161
- [Background] Selya AS, Rose JS, Dierker LC, Hedeker D, Mermelstein RJ. A Practical Guide to Calculating Cohen's f(2), a Measure of Local Effect Size, from PROC MIXED. Front Psychol. 2012 Apr 17;3:111. doi: 10.3389/fpsyg.2012.00111. eCollection 2012. PMID 22529829
- [Background] Dong Z, Zhu Y, Du H, Wang J, Zeng X, Tao X, Yang T, Wang J, Deng M, Liu J, Wu L, Yu H. The effectiveness of a computer-aided system in improving the detection rate of gastric neoplasm and early gastric cancer: study protocol for a multi-centre, randomized controlled trial. Trials. 2023 May 11;24(1):323. doi: 10.1186/s13063-023-07346-5. PMID 37170280
- [Background] Boonstra AM, Stewart RE, Koke AJ, Oosterwijk RF, Swaan JL, Schreurs KM, Schiphorst Preuper HR. Cut-Off Points for Mild, Moderate, and Severe Pain on the Numeric Rating Scale for Pain in Patients with Chronic Musculoskeletal Pain: Variability and Influence of Sex and Catastrophizing. Front Psychol. 2016 Sep 30;7:1466. doi: 10.3389/fpsyg.2016.01466. eCollection 2016. PMID 27746750
- [Background] Cleland JA, Childs JD, Whitman JM. Psychometric properties of the Neck Disability Index and Numeric Pain Rating Scale in patients with mechanical neck pain. Arch Phys Med Rehabil. 2008 Jan;89(1):69-74. doi: 10.1016/j.apmr.2007.08.126. PMID 18164333
- [Background] Sim J, Jordan K, Lewis M, Hill J, Hay EM, Dziedzic K. Sensitivity to change and internal consistency of the Northwick Park Neck Pain Questionnaire and derivation of a minimal clinically important difference. Clin J Pain. 2006 Nov-Dec;22(9):820-6. doi: 10.1097/01.ajp.0000210937.58439.39. PMID 17057565
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714